CLINICAL TRIAL: NCT02952365
Title: A Prospective Evaluation of Tissue Sealant to Prevent Epithelial Ingrowth in Repeat LASIK Surgery
Brief Title: Tissue Sealant Use in LASIK Enhancement Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Edward E. Manche, Principal Investigator, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: IRB-38495
Record Dates: First submitted 2016-10-27; First posted 2016-11-02 (Estimated); Results first posted 2021-12-14 (Actual); Last update posted 2021-12-14 (Actual); Status verified 2021-11

CONDITIONS: Epithelial Ingrowth
Keywords: LASIK, Ingrowth, Tissue sealant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Eyes undergoing LASIK enhancement (Other): Eyes undergoing LASIK enhancement will have tissue sealant applied to the eye to prevent epithelial ingrowth
  Interventions: Drug: Tissue sealant

INTERVENTIONS:
Drug: Tissue sealant — Application of tissue sealant on eyes undergoing LASIK enhancement
  Other Names: ReSure sealant

SUMMARY:
The purpose of the study is to evaluate the use of prophylactic tissue sealant to prevent epithelial ingrowth from gaining access under a LASIK flap with repeat LASIK surgery

DETAILED DESCRIPTION:
Participants will have a comprehensive eye examination once they express an interest in the study. This includes a slit lamp examination of the front of the eye and a dilated fundoscopic examination of the back of the eye. If there is any pathology noted that would exclude the participant from the study, then the participant will be informed and given an appropriate referral. If the participant is deemed appropriate for the study after a comprehensive examination included computerized videokeratography, then they can be enrolled. The participant will undergo LASIK flap lift eye surgery.

Tissue sealant will be applied at to the edge of the LASIK flap at the conclusion of the surgery. A bandage contact lens will also be placed. The bandage contact lens is used in the usual and customary fashion as in non-study LASIK flap lift surgery.

The participants will be seen on the day of surgery, post op day one, one month, and three months. The participant will receive topical antibiotics in each eye for one week following the procedure. The participant will receive pred forte 1% ophthalmic drops for one week after treatment. The participant will also receive vigamox ophthalmic drops for seven days after treatment. All of this is within the usual and customary standard of care for the treatment of participants undergoing LASIK surgery.

ELIGIBILITY:
Inclusion Criteria:

* Subjects age 21 and older
* Subjects with healthy eyes
* Subjects who have previously undergone LASIK surgery
* Subjects with residual refractive error.

Exclusion Criteria:

* Subjects under the age of 21.
* Subjects with excessively thin corneas.
* Subjects with topographic evidence of keratoconus.
* Subjects with ectatic eye disorders.
* Subjects with autoimmune diseases.
* Subjects who are pregnant or nursing.

Ages: 21 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2016-10-01 (Actual); Primary Completion 2017-05-22 (Actual); Study Completion 2017-05-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Edward E Manche, MD, Principal Investigator — Stanford University
Locations (1):
- Byers Eye Institute at Stanford, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: Eyes
Period: Overall Study
Arm/Group | Eyes Undergoing LASIK Enhancement
Started | 2; 2 Eyes
Completed | 2; 2 Eyes
Not Completed | 0; 0 Eyes

BASELINE CHARACTERISTICS:
Units Other Than Participants: Eyes
Arm/Group | Eyes Undergoing LASIK Enhancement
Number analyzed (Participants) | 2
Number analyzed (Eyes) | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 2

OUTCOME MEASURES:

1. Primary Outcome: Slit Lamp Examination for Presence of Epithelial Ingrowth Under LASIK Flap
Description: The number of eyes that developed epithelial ingrowth under LASIK flap
Time Frame: At post-operative month 3
Measure: Count of Units; unit: Eyes
Units Other Than Participants: Eyes
Arm/Group | Eyes Undergoing LASIK Enhancement
Number analyzed (Participants) | 2
Number analyzed (Eyes) | 2
Eyes | 0

2. Secondary Outcome: Change in Refraction
Description: Number of eyes within 0.5 diopters of the intended correction
Time Frame: At post-operative month 3
Measure: Count of Units; unit: Eyes
Units Other Than Participants: Eyes
Arm/Group | Eyes Undergoing LASIK Enhancement
Number analyzed (Participants) | 2
Number analyzed (Eyes) | 2
Eyes | 2

3. Secondary Outcome: Best-corrected Visual Acuity
Description: Number of eyes losing 2 or more lines of corrected distance visual acuity measured by ETDRS testing charts
Time Frame: At post-operative month 3
Measure: Count of Units; unit: Eyes
Units Other Than Participants: Eyes
Arm/Group | Eyes Undergoing LASIK Enhancement
Number analyzed (Participants) | 2
Number analyzed (Eyes) | 2
Eyes | 0

4. Secondary Outcome: Uncorrected Visual Acuity
Description: Number of eyes with an uncorrected visual acuity of 20/20 at 12 months measured using ETDRS testing charts
Time Frame: At post-operative month 3
Measure: Count of Units; unit: Eyes
Units Other Than Participants: Eyes
Arm/Group | Eyes Undergoing LASIK Enhancement
Number analyzed (Participants) | 2
Number analyzed (Eyes) | 2
Eyes | 2

ADVERSE EVENTS:
Time Frame: 3 months
Description: Data on all serious and non-serious Adverse Events experienced by participants were collected, irrespective of the event's relation to the treated eye.
Arm/Group | Eyes Undergoing LASIK Enhancement
All-Cause Mortality (participants affected / at risk) | 0/2
Serious Adverse Events (participants affected / at risk) | 0/2
Other Adverse Events (participants affected / at risk) | 0/2

LIMITATIONS AND CAVEATS:
The study did not meet its planned enrollment number

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-09-20): https://cdn.clinicaltrials.gov/large-docs/65/NCT02952365/Prot_SAP_000.pdf